CLINICAL TRIAL: NCT07184333
Title: Interprofessional Education and Connected Care: A Home-Based Digital-Integrated Frailty Management Programme for Older Adults With Mild Impairments
Brief Title: Interprofessional Education Programme for Nursing and Physiotherapy Students Providing Home-Based Care to Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Agnes LAI Yuen Kwan, Associate Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HE-T&L2025/03
Record Dates: First submitted 2025-08-27; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Frailty at Older Adults
Keywords: Interprofessional education; home-based care; frailty; interprofessional collaboration; older adults; nursing; physiotherapy; student
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interprofessional Education with Digital Case Management Platform (Experimental): This arm includes nursing and physiotherapy student participants who receive an interprofessional education intervention involving structured training workshops, supervised home visits, and use of a tablet-based digital case management platform. The intervention aims to enhance students' clinical competencies, digital health literacy, and interprofessional collaboration skills in the context of delivering home-based care to community-dwelling older adult participants with mild impairments. The older adult participants, referred through a local social service agency, receive health assessments, education, and personalised care planning during structured home visits conducted by student teams. The intervention also incorporates the use of mobile health messages and wearable devices to support follow-up care and engagement.
  Interventions: Behavioral: Interprofessional Education with Digital Case Management for Home-Based Elder Care

INTERVENTIONS:
Behavioral: Interprofessional Education with Digital Case Management for Home-Based Elder Care — A structured interprofessional education programme for nursing and physiotherapy students that includes: (1) a 3-hour workshop on frailty assessment, digital case documentation, and care planning; (2) a 30-minute orientation on home visit safety and communication; (3) supervised home visits to older adult participants involving health and fitness assessments, medication support, and health education; (4) use of a tablet-based digital case management platform for collaborative care documentation; and (5) a 4-week follow-up with personalised mobile health messages and a final home visit. The intervention aims to enhance students' clinical, collaborative, and digital competencies in community-based elder care.

SUMMARY:
The goal of this mixed-methods research is to investigate the impact of interprofessional education on the professional development and clinical skills of nursing and physiotherapy students who provide home-based care to older adults in Hong Kong. The main questions it aims to answer are:

1. Is an interprofessional home-based digital frailty management program feasible for training nursing and physiotherapy students ?
2. Can the training enhance students' skills in providing holistic, home-based care, interprofessional teamwork and communication?
3. Can the training improve elderly health awareness, behavior, and outcomes?

The study will involve 50 students from Hong Kong Metropolitan University, including nursing and physiotherapy students in clinical placement courses. Approximately 100 older adults with mild health conditions, living in home-based community settings, will take part as care recipients.

Students will:

1. Attend a training programme delivered by healthcare professionals, including nurses, physiotherapists, and social workers.
2. Carry out supervised home visits in pairs, working directly with older adults to assess their needs, provide health education, and support healthy lifestyle changes.
3. Use a tablet-based digital platform to record care plans, share information, and follow up with participants.

DETAILED DESCRIPTION:
Background: The global ageing population has created a growing demand for healthcare services, particularly for older adults with chronic conditions and complex care needs. In Hong Kong, home-based community care services are delivered through government-NGO partnerships, allowing older adults to stay within their communities while enhancing their quality of life. Interprofessional education (IPE), which involves collaborative learning among students from different health and social care professions, is a proven approach to fostering teamwork, effective communication, and patient-centred care. However, IPE programmes in Hong Kong are often classroom-based, with limited opportunities for real-world application in community care settings.

Objectives: The project aims to assess the feasibility of an interprofessional home-based digital frailty management program that integrates professional education and community services, enhancing students' skills in providing holistic, home-based care, interprofessional teamwork and communication, and improving elderly health awareness, behavior, and outcomes.

Methods: With strong academic-community partnerships, 50 nursing and physiotherapy students will enrol in a 3-month clinical placement programme. Prior to the clinical placement, students will participate in a two-session training workshop, conducted by a multidisciplinary team including nurses, physiotherapists, and social workers. During the placement, students will conduct supervised home visits to approximately 60 families, involving around 100 older adults with mild impairments, focusing on the elderly's frailty, including brief health, frailty, and home safety assessments and education on medication adherence, healthy living habits, and the use of "HA Go" and instant messaging. Students will use a digital case management and handover platform to enter all elderly information, issues, management plans, and actions for handover and follow-up. For each visit, at least one of the team members will accompany students to conduct the visit. After the first home visit, Students will also deliver booster e-health mobile messages (twice a week for a month). One month after the first home visit, the second home visit to these elderly will be conducted by students to assess their health-related behaviour changes and improvement in home safety. Four levels of evalauation framework will be used to assess students' satisfaction with the program (reaction), changes in perceived skills and knowledge, or attitudes after program completion (competency), and the extent to which changes in professional behaviour in actual clinical work (clinical practice), changes in elderly's health-related behaviour (health care outcomes). The first three levels will be conducted for students through questionnaire surveys and qualitative interviews at three time points: prior to the training (T1), immediately after the completion of clinical placement (T2), and three months post-training (T3). The fourth level will be conducted for the elderly at the first home visit and one month after the first home visit. Findings will be disseminated through academic publications and conference presentations.

Expected Impacts: This programme will integrate student learning with community service, benefiting students, communities, academia, and policy. For students, it will enhance students' skills in interprofessional collaboration, communication, and holistic, person-centered care while building confidence through hands-on experience with digital case management platforms. The digital case management handover platform provides hands-on practice in case handover, management, action planning, and follow-up for elderly care, with potential applications in other programs or courses. For communities, it will promote healthier aging by improving health awareness, enabling early detection of concerns, and enhancing care services through regular student and teacher interactions. In academia and policy, it will provide evidence to guide educational approaches, support the adoption of digital tools, and promotes innovative healthcare education.

ELIGIBILITY:
Students

Inclusion criteria:

* Aged 18 years or above.
* Nursing students: Year 3 Higher Diploma in Nursing students at HKMU enrolled in NURS N222C Clinical Practicum. OR Physiotherapy students: Year 3 and Year 4 Bachelor of Science (Hons) in Physiotherapy students at HKMU enrolled in PHSI N212F Clinical Practicum II.
* Able to read Chinese and English, and speak Cantonese.
* Willing to participate in the training workshop and conduct home-based intervention.

Older Adults

Inclusion criteria:

* Aged 60 years or above.
* Service users of AKA.
* Mild impairments (non-bedbound, physically capable of participating in simple exercises).
* Able to read Chinese and/communicate in Cantonese.
* Willing to participate in health surveys, home visits, and follow-ups, and to receive and respond to text messages.
* Must own a smartphone and know how to use it.

Students

Exclusion criteria:

* Unwilling to provide consent.
* Cannot read Chinese or speak Cantonese.

Older adults

Exclusion criteria:

* Not a registered service user from AKA.
* Unwilling to provide consent.
* Cannot read Chinese or speak Cantonese.
* Unwilling to participate in the interventions conducted by students.
* Severe communication impairments.
* Do not own a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in students' satisfaction and self-confidence in learning | Immediately after the training workshop; immediately after the follow-up home visit (4-week); three months after the training workshop
  This outcome will assess students' satisfaction with the program and their self-confidence in mastering the learned knowledge and skills. The 10-item Modified Student Satisfaction and Self-Confidence in Learning Scale includes two subscales: satisfaction with the program (items 1-5) and self-confidence in learning (items 6-10). Each item is rated on a 5-point Likert scale from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Subscale scores are summed, with higher scores indicating greater satisfaction or confidence.

SECONDARY OUTCOMES:
Changes in students' clinical practice in team and patient interaction | Prior to the training workshop; immediately after the follow-up home visit (4-week); three months after the training workshop
  This outcome assesses changes in students' clinical practice during interprofessional education placements, focusing on interactions with both team members and patients. The 8-item Clinical Practice on Team and Patient Interaction Scale includes two subscales: Team Interaction (items 1-4) evaluates collaboration, communication, role understanding, and decision-making; Patient Interaction (items 5-8) assesses rapport-building, cultural sensitivity, health education, and professionalism. Each item is rated on a 5-point Likert scale from 1 ("Strongly Disagree" or "Not at all effective") to 5 ("Strongly Agree" or "Extremely effective"). Scores are summed, with higher scores indicating more effective clinical interactions.
Changes in students' perceptions of interprofessional clinical education and collaborative practice | Immediately after the training workshop; immediately after the follow-up home visit (4-week); three months after the training workshop
  This outcome evaluates students' perceptions of interprofessional teamwork, roles and responsibilities, and patient outcomes following participation in the interprofessional education program. The 10-item Perceptions of Interprofessional Clinical Education (Revised) survey is used, with items divided into three domains: teamwork, roles/responsibilities, and patient outcomes. Each item is rated on a 5-point Likert scale from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). Higher total and subscale scores indicate more positive perceptions of interprofessional learning and collaborative practice.
Students' perceived usefulness and ease of use of the digital handover platform | Immediately after the follow-up home visit (4-week)
  This outcome assesses students' acceptance of the digital case management handover platform using the 12-item Technology Acceptance Model (Version 4). The instrument includes two subscales: Perceived Usefulness (items 1-6) evaluates how the platform supports productivity, job performance, and effectiveness, while Ease of Use (items 7-12) measures usability, clarity, control, and flexibility. Items are rated on a 7-point Likert scale from 1 ("Extremely Disagree") to 7 ("Extremely Agree"). Higher total and subscale scores indicate more favorable perceptions of the platform's usability and usefulness.
Changes in anxiety and depression symptoms among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  This outcome evaluates changes in older adults' mental health by measuring symptoms of anxiety and depression using the 4-item Patient Health Questionnaire-4 (PHQ-4). The tool includes two items for anxiety and two for depression. Each item is rated on a 4-point scale from 0 ("Not at all") to 3 ("Nearly every day"), producing a total score ranging from 0 to 12. Scores are interpreted as follows: normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Higher scores indicate greater psychological distress.
Changes in sleep quality among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  This outcome assesses changes in sleep quality and insomnia symptoms among older adults using the Insomnia Severity Index (ISI). The ISI is a 7-item self-reported questionnaire evaluating the severity of sleep-onset and sleep-maintenance difficulties, satisfaction with sleep, and the impact of insomnia on daily functioning. Each item is rated on a 5-point Likert scale, with total scores ranging from 0 to 28. Scores are interpreted as follows: no clinically significant insomnia (0-7), subthreshold insomnia (8-14), moderate clinical insomnia (15-21), and severe clinical insomnia (22-28). Higher scores indicate greater insomnia severity.
Changes in sense of loneliness among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  This outcome evaluates the emotional and social loneliness of older adults using the De Jong Gierveld Loneliness Scale, a validated 6-item instrument. The scale includes two subscales: Emotional Loneliness (EL) (items 1-3) and Social Loneliness (SL) (items 4-6). Responses are scored differently based on item phrasing: for negatively worded items (1-3), "Yes" and "More or less" are scored as 1, and "No" as 0; for positively worded items (4-6), "Yes" is scored as 0, "More or less" as 1, and "No" as 1. Total scores range from 0 (least lonely) to 6 (most lonely). Higher scores reflect greater loneliness.
Changes in physical activity levels among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  This outcome evaluates older adults' physical activity levels using the International Physical Activity Questionnaire - Short Version (IPAQ-SF). This 7-item self-reported tool captures the frequency (days per week) and duration (minutes per day) of physical activity performed at three intensity levels: vigorous activity, moderate activity, and walking, as well as sedentary behavior (sitting time). Participant responses are converted into Metabolic Equivalent Task (MET)-minutes per week, providing a standardized estimate of overall physical activity. Higher MET scores indicate greater physical activity levels.
Changes in happiness among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  Older adults subjectively report their general happiness using an 11-point Likert scale (0 = "not at all" to 10 = "totally"), responding to a question: "I feel happy in general".
Changes in frailty status among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  This outcome evaluates frailty using the Fried's Frailty Phenotype Tool, a validated and widely used assessment consisting of five criteria:
  Unintentional weight loss: ≥4.5 kg or ≥5% of body weight lost in the past year Exhaustion: Self-reported fatigue on ≥3 days per week Low physical activity: No moderate-intensity activity for at least 10 minutes per day Slow walking speed: Gait speed below threshold based on height and gender Weak grip strength: Grip strength below threshold based on gender and BMI
  Each criterion is scored as 1 (present) or 0 (absent). The total score ranges from 0 to 5 and classifies individuals as:
  Robust: 0 criteria Pre-frail: 1-2 criteria Frail: ≥3 criteria The tool combines objective measures (e.g., walking speed, grip strength) and subjective responses (e.g., fatigue), and is highly predictive of adverse health outcomes in older adults.
Changes in confidence in managing chronic illness among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  This outcome measures self-efficacy in managing chronic disease using the Self-Efficacy for Managing Chronic Disease Scale. This 6-item questionnaire asks older adults to rate their confidence in performing various self-management activities despite their chronic condition. Each item is scored on a 10-point Likert scale ranging from 1 ("not at all confident") to 10 ("totally confident"). The final score is calculated as the mean of at least 4 items, allowing up to 2 missing responses. Higher scores indicate greater confidence in managing one's chronic illness.
Changes in medication adherence among older adults | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  Morisky Medication Adherence Scale (MMAS-8) is used to assess patient adherence to prescribed medications for chronic conditions. The scoring involves summing responses from eight items, where seven are yes/no ("no" answers receive a score of 1 point) and the eighth uses a 5-point Likert scale (never =1, once in a while =0.75, sometimes =0.5, usually =0.25, and all the time =0), with a total score ranging from 0 to 8. Higher scores indicate better medication adherence. Adherence is categorized as Low (score <6), Medium (score 6 to <8), and High (score = 8).
Changes in Polypharmacy Risk | During the first home visit (T1, baseline); during the follow-up home visit (T2, 4-week)
  Polypharmacy Risk is assessed by three items: 1) Are you regularly taking five or more medications? 2) Are you taking any of the following medications? (Anticoagulants, diabetes medications, psychiatric and neurological medications); 3) Have you changed your medications in the past eight weeks?. A response of yes for any items indicates a high risk.
Wrist-worn digital watch measured step counts | Immediately after the first home visit (T1, baseline); Immediately after the follow-up home visit (T2, 4-week)
  Wrist-worn digital watch measured daily step counts (total number of steps per day)
Wrist-worn digital watch measured sleep time | Immediately after the first home visit (T1, baseline); Immediately after the follow-up home visit (T2, 4-week)
  Wrist-worn digital watch measured daily sleep time (duration of sleep per day, hours)

OTHER OUTCOMES:
Qualitative feedback: students' perceptions of interprofessional training and its impact on IPE competency | Within 1 month after the completion of the follow-up home visits (4-week)
  This outcome involves qualitative data collection through focus group interviews with approximately 20 students (nursing and physiotherapy). Participants will be selected using purposive sampling to ensure diversity in IPE experience. The final number of participants will be determined based on data saturation, defined as the point when no new themes emerge.
  The interviews will explore:
  Perceptions of the interprofessional education (IPE) training workshops Perceived impact on IPE core competencies (e.g., collaboration, communication, role clarity) Reflections on interprofessional home visit experiences This qualitative approach aims to provide contextual understanding and deeper insights into the educational intervention's effectiveness, complementing the quantitative evaluation of IPE outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- School of Nursing & Health Sciences, Hong Kong Metropolitan University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The trial does not include provisions for data sharing due to privacy concerns and absence of participant consent for secondary data use.